CLINICAL TRIAL: NCT06545968
Title: Retention Through mHealth for Adolescents and Young Adults With HIV in Care
Brief Title: A Social Media Intervention to Improve Retention in Care for Adolescents and Young Adults With HIV in Uganda
Acronym: REMAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUST-2024-06-14; K43TW012640 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Behavior
Keywords: Adolescents and young adults; HIV; mHealth; Retention in care
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The proposed project is a mixed-methods prospective cohort study of adolescents and young adults with HIV, clinic counsellors. The study will design and test a social media mHealth intervention to improve retention in care for adolescents and young adults with HIV.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): These are the participants who will be randomised to receive the intervention at the start of the study.
  Interventions: Behavioral: A social media based intervention
- Wait list control arm (No Intervention): These are participants who will not receive the intervention initially, but will move to the intervention arm after 6 months of follow-up

INTERVENTIONS:
Behavioral: A social media based intervention — WatsApp-based modules to influence retention in care behaviour
  Arms: Intervention arm

SUMMARY:
Adolescents and young adults with HIV (AYWH) aged 15- 24 years are the fastest-growing population of people living with HIV worldwide. AYWH have worse outcomes along the HIV continuum of care than adults with HIV; HIV/AIDS is the second leading cause of mortality and the fourth leading cause of disability among AYWH worldwide. This study will develop a youth-friendly, mobile health (mHealth) intervention to improve retention in care that has the potential to improve AIDS-related mortality and morbidity among AYWH and decrease onward new transmission, thus contributing towards ending the HIV/AIDS pandemic.

DETAILED DESCRIPTION:
Background: Of the adolescents and young adults with HIV (AYWH) who initiate in care, only about 50% remain in care at 12 months; in 2020, AYWH recorded a 50% increase in AIDS-related mortality. These poor clinical outcomes among AYWH are multi-factorial and largely influenced by their neurodevelopmental stage and differ by route of infection. Current interventions to retain AYWH in care are ineffective and do not address the neurodevelopmental issues of AYWH. Social media-based mHealth interventions may offer flexible and attractive features to AYWH to help overcome these barriers. Candidate: The goal of the proposed K43 Emerging Global Leader Award is to support The investigator's research training to attain independence as a clinician-scientist focused on improving treatment and care for AYWH in low resourced settings. The investigator is currently a research fellow at Mbarara University of Science and Technology, Uganda. The proposed study will enable training in three areas: 1) Qualitative research skills, including design, data collection, analysis and interpretation; 2) Behavioural science skills to better understand influences of adolescent behaviour and implications for mHealth-based intervention development and deployment; 3) Skills in statistical methods for clinical trials to conduct clinical trials and longitudinal data analysis. This application builds on The investigator's current clinical experience and background in epidemiology, as well as ongoing formative work in mHealth intervention development and a highly supportive, multidisciplinary team of mentors. Research: The research goals of this proposal are to develop and test a psychosocial social media-based mHealth intervention to improve retention in care of AYWH attain viral suppression, therefore decreasing AIDS-related mortality and preventing onward HIV transmission. The investigator will identify the HIV knowledge gaps, experiences, and challenges among AYWH who are new or re-engaging in HIV care, characterizing these factors by route of infection (i.e., perinatal vs non-perinatal) among AYWH in resource limited populations.

ELIGIBILITY:
The eligibility criteria is as follows:

For adolescents and young adults with HIV (AYWH)

1. AYWH who are aged 15-24
2. AYWH who are new to care (less than or equal to one month in care), or who are re-engaging in care after being lost to follow up for greater or equal to six months.
3. Fluent in English or Runyankole (the local language)
4. For aim 3, AYWH who have access (own or shared) to a smartphone

Exclusion criteria for AYWH 1) Inability to provide consent

For counsellors Inclusion criteria

1. Clinic counsellors who are ≥18 years
2. Clinic counsellors who have worked at the HIV clinic for ≥ 1 year

Exclusion criteria

1) Inability to provide consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary intervention outcome will be the acceptability, feasibility of the intervention. | 12 months
  Acceptability will be measured using the Acceptability of Intervention Measure (AIM) and will be considered acceptable if ≥70% (35/50) of intervention participants rate all 4 items on the AIM (a 5-point Likert scale) as "agree" or higher.
  The intervention will be considered feasible if ≥70% (35/50) of intervention participants rate all 4 items on the Feasibility of Intervention Measure (FIM), (a 5-point Likert scale) as "agree" or higher.

SECONDARY OUTCOMES:
Retention | 12 months
  The secondary outcome of the intervention will be retention in care, which will be assessed at the end of 12 months. This will be defined as the proportion of participants active in care (i.e have not missed a scheduled appointment in the last 12 months) The investigators will compare the proportion of participants actively engaged in care in the immediate intervention and the deferred intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Adong, MMed, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT06545968/Prot_SAP_000.pdf